CLINICAL TRIAL: NCT06449846
Title: Compare the Accuracy of Circulating Tumor DNA Longitudinal Monitoring Minimal Residual Disease and Microvascular Invasion Result in Predicting Postoperative Recurrence of Hepatocellular Carcinoma
Brief Title: Compare the Accuracy of ctDNA-MRD and MVI Result in Predicting Postoperative Recurrence of Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KY-094-02
Record Dates: First submitted 2024-04-30; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma Resectable; Surgery; Recurrence
Keywords: Hepatocellular Carcinoma; Circulating Tumor DNA; Minimal Residual Disease; Microvascular Invasion
MeSH Terms: conditions — Recurrence; Carcinoma, Hepatocellular; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with hepatocellular carcinoma: Patient with hepatocellular carcinoma who can undergo radical resection
  Interventions: Diagnostic Test: circulating tumor cell DNA detection

INTERVENTIONS:
Diagnostic Test: circulating tumor cell DNA detection — circulating tumor DNA blood sample and tissue specimen for circulating tumor DNA will be done to patient with hepatocellular carcinoma

SUMMARY:
The aim of this study was to compare the accuracy of ctDNA-MRD longitudinal surveillance model and internationally accepted pathological MVI results in predicting recurrence after radical hepatectomy. At the same time, to explore the relationship among the two methods of predicting recurrence of hepatocellular carcinoma, postoperative adjuvant therapy and postoperative recurrence, this study further confirmed the effectiveness of ctDNA-MRD longitudinal monitoring model in monitoring postoperative recurrence of hepatocellular carcinoma and guiding treatment.

DETAILED DESCRIPTION:
The recurrence rate of hepatocellular carcinoma (HCC) after radical hepatectomy is high, and there is no universally accepted adjuvant therapy to prevent recurrence of liver cancer at present.The high-risk recurrent population can not be accurately and dynamically located. The results showed that minimal residual disease (MRD) was the root of recurrence of HCC, and the results of MRD were the important indicator of adjuvant therapy. Our previous research confirmed that the circulating tumor DNA (ctDNA)-MRD monitoring model can accurately predict the recurrence of HCC, which provides important evidence for the application of MRD in predicting the recurrence of early HCC. It was also found in the retrospective analysis that the patients with ctDNA positive after radical hepatectomy were treated with targeted therapy and other comprehensive therapies, while ctDNA converting to negative, the tumor-free survival was significantly prolonged.

Microvascular invasion (MVI) is a pathological concept, which refers to the nests of cancer cells in the lumen of small blood vessels under the microscope, the results of MVI can be obtained by pathological examination of the tumor tissue after hepatectomy. MVI is common in HCC and is associated with early recurrence and decreased survival. MVI is an important determinant of survival after radical hepatectomy, the grade (severity) of MVI is generally associated with tumor stage and the rate of liver cancer disease progression, which has been widely studied and recognized internationally.

The aim of this study was to compare the accuracy of ctDNA-MRD longitudinal surveillance model and internationally accepted pathological MVI results in predicting recurrence after radical hepatectomy. At the same time, to explore the relationship among the two methods of predicting recurrence of hepatocellular carcinoma, postoperative adjuvant therapy and postoperative recurrence, this study further confirmed the effectiveness of ctDNA-MRD longitudinal monitoring model in monitoring postoperative recurrence of hepatocellular carcinoma and guiding treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-75 years;
2. Preoperative imaging examination diagnosed hepatocellular carcinoma (BCLC) stage 0/ stage A/stage B, eligible for radical surgery;
3. ECOG physical status score is 0-1;
4. Child-Pugh score is 5-6 points (Level A);
5. Not received any anti-tumor therapy;
6. Laboratory tests were at normal levels within 7 days before enrollment.

Exclusion Criteria:

1. Patient can't provide blood samples for ctDNA testing;
2. Patient with two or more types of tumors at the same time;
3. Non-primary liver lesions;
4. Pregnant or lactating women;
5. Patient with a history of other malignant tumors within the past 5 years or at the same time, except cured skin basal cell carcinoma, cervical carcinoma in situ and thyroid papillary carcinoma;
6. Patient with serious heart disease;
7. Other conditions deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with hepatocellular carcinoma who can undergo radical surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The ROC curve of two methods are obtained according to the results of recurrence prediction 2 years after hepatectomy，and the primary outcome measure is the area under the ROC curve (AUC value) for two methods | 2 years
  The receiver operating characteristic curve (ROC) is made according to the recurrence of the patients after operation, and the accuracy of ctDNA-MRD longitudinal monitoring model and pathological MVI results are judged by comparing the area under the ROC curve (AUC value)

SECONDARY OUTCOMES:
2-year recurrence-free survival rate | 2 years
  percentage of recurrence-free survival 2 years after surgery

OTHER OUTCOMES:
1-year recurrence-free survival rate | 1 years
  percentage of recurrence-free survival 1 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mingxin Pan, Prof., Principal Investigator — Southern Medical University
Locations (4):
- China (4):
  - Shunde Hospital of Southern Medical University, Foshan, Guangdong
  - The Sixth Affiliated Hospital of South China University of Technology, Foshan, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guanzhou, Guangdong